CLINICAL TRIAL: NCT05807997
Title: Patients Who Were Not Admitted to the Intensive Care Unit: Characteristics and Clinical Outcomes. Retrospective Study
Status: Recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: 0075-23-MMC
Record Dates: First submitted 2023-03-16; First posted 2023-04-11 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Refusal of ICU Admission

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Refusal of ICU admission. — patients aged 18--99 who were presented to the general intensive care unit from January 2018 to the end of December 2023 and were not admitted.

SUMMARY:
There is extensive medical literature supporting the contribution of intensive care physicians to improvement of clinical outcomes in patients treated in an intensive care unit (1-3). There are many reasons for this contribution, including adherence to evidence-based medical protocols, as well as collaboration between different medical specialties in patient care (4-7). Over the years, several criteria have been formulated for the admission of patients to intensive care (8) according to their medical condition, but there are other factors that influence the decision whether to admit patients to intensive care, not necessarily medical ones, such as the availability of beds in the unit and the availability of medical and nursing staff.

There are several studies that examined the characteristics and clinical outcomes of patients who were not admitted to the intensive care unit, for medical or paramedical reasons (9). We would like to retrospectively examine all patients in the last 5 years who were presented for admission to general intensive care from various departments in our institution but were not admitted, to characterize the reasons why they were not admitted, the clinical characteristics of the patients and their clinical outcomes.

Objectives:

Main objective:

To characterize the clinical outcomes of the patients who were presented for admission to general intensive care but were not admitted in the last 5 years.

Secondary objectives:

To characterize the reasons why the patients were not admitted - medical and paramedical, and to examine the clinical characteristics of these patients (age, sex, background diseases and current disease.).

Design and methods:

Study design:

This is a retrospective study based on data collection.

Methods and materials:

Collecting information from computer systems regarding the patients who were presented by the various departments at the Meir Hospital in Kfar Saba for admission to the general intensive care unit and were not admitted, starting from the beginning of January 2018 until the beginning of January 2023. These are about 1000 patients. After the end of data collection in the study, the data will be typed anonymously into a dedicated Excel file. The patients will be identified according to the patient number in the study and the case number, without specifying identifying details.

Inclusion criteria:

All patients aged 18--99 who were presented to the general intensive care unit from January 2018 to the end of December 2023 and were not admitted.

Data collection:

The research will be conducted in the format of observational data collection from the patient files and from computerized systems (Camelion system and iMDsoft software).

The data collected in the study will be exposed to the research team only as long as the actual data collection is carried out. After the end of data collection in the study, the data will be typed anonymously into a dedicated Excel file. The patients will be identified according to the patient number in the study and the case number, without specifying identifying details.

The data to be collected: age, sex, underlying diseases, regular medications, duration of hospitalization, need for ventilation, number of days of ventilation, mortality within 28 days, APACHE-2 score, SOFA score, lactate level, need for pressors, need for dialysis or other RRT, The reasons for not being admitted to the intensive care unit.

Size of the research group: about 1000 patients - this is the estimated number of patients in the time period detailed above.

The method of processing the results: all the demographic and in-hospital indicators will be tested statistically by a certified statistician depending on the type of data.

ELIGIBILITY:
Inclusion Criteria:All patients aged 18--99 who were presented to the general intensive care unit from January 2018 to the end of December 2023 and were not admitted.

-

Exclusion Criteria:None

-

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients aged 18--99 who were presented to the general intensive care unit from January 2018 to the end of December 2023 and were not admitted.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
28-day mortality among unadmitted patients | 5 years
  To assess 28-day mortality of the patients who were presented for admission to general intensive care but were not admitted

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No